CLINICAL TRIAL: NCT01934582
Title: A Pharmacokinetic Substudy of Subjects Transitioning From Twice Daily to Three Times Daily Dosing of UT-15C SR (Treprostinil Diethanolamine) in the TDE-PH-304 Protocol
Brief Title: A Pharmacokinetic Substudy of the TDE-PH-304 Protocol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TDE-PH-309; TDE-PH-304
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Results first posted 2016-10-27 (Estimated); Last update posted 2024-01-03 (Actual); Status verified 2016-09

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label extension (Experimental)
  Interventions: Drug: UT-15C SR; Drug: treprostinil diethanolamine

INTERVENTIONS:
Drug: UT-15C SR
Drug: treprostinil diethanolamine — Open label study drug.
  Other Names: UT-15C Sustained Release (SR)

SUMMARY:
A sub-study to the TDE-PH-304 protocol to assess the pharmacokinetics of patients transitioning from a twice daily dosing regimen of oral treprostinil to a three times daily dosing regimen.

DETAILED DESCRIPTION:
As noted above in "Brief Summary".

ELIGIBILITY:
Inclusion Criteria:

1) Only subjects who are eligible for and have entered into Protocol TDE-PH-304 may participate in this substudy.

Exclusion Criteria:

1. The subject must voluntarily give informed consent to participate in the substudy.
2. No dose changes to study drug are made within 5 days of the pharmacokinetic (PK)substudy visits.
3. No additions or deletions to concurrent medications are made within 7 days of the pharmacokinetic substudy visit. Note: changes to diuretics and/or anticoagulants are permitted.
4. The preceding evening dose of study drug should have been taken 9 to 13 hours prior to the BID dose and 6-10 hours prior to the TID morning dose of study drug to ensure a trough level of study drug for PK sampling.
5. Subject dosing of study drug on the day of PK sampling must be observed in the clinic by study personnel.
6. Subject has not experienced a significant loss of blood (> 450 mL) within the last 6 weeks of the pharmacokinetic substudy visit.
7. The subject must not be receiving any CYP 2C8 inducers or inhibitors

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R White, MD, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label Extension PK Population: The PK population included all subjects enrolled in the PK substudy having met the study criteria who received at least 1 treatment of open-label treprostinil diethanolamine.
Period: Overall Study
Arm/Group | Open-label Extension PK Population
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Open-label Extension PK Population: The PK population included all subjects enrolled in the PK substudy having met the study criteria, who had sufficient treprostinil concentration-time data to derive noncompartmental PK parameters for at least 1 treatment of open-label treprostinil diethanolamine.
Arm/Group | Open-label Extension PK Population
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: years] | 60.6 [38 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Pharmacokinetics (Mean AM Dose) in Subjects During Twice Daily (BID) Dosing (up to 14 Days Prior to Transitioning to Three Times Daily [TID] Dosing Regimen at PK Visit 1) and up to 35 Days After Transitioning to TID Dosing (at PK Visit 2).
Description: The PK sampling occurred over a 12-hour period in subjects during BID dosing (PK Visit 1) and during TID dosing (PK Visit 2). Prior to each PK sampling day, subjects must have been receiving a stable dose for at least 5 days.
Time Frame: Up to 14 days prior to transitioning to TID dosing regimen (PK Visit 1) and up to 35 days after transitioning to TID dosing regiment (PK Visit 2)
Measure: Mean (Full Range); unit: mg
Groups:
- PK Visit 1: UT-15C SR (treprostinil diethanolamine) BID
- PK Visit 2: UT-15C SR (treprostinil diethanolamine) TID
Arm/Group | PK Visit 1 | PK Visit 2
Number analyzed (Participants) | 13 | 13
mg | 8.12 [2.00 to 17.5] | 6.75 [1.25 to 15.0]

2. Primary Outcome: To Assess the Pharmacokinetics (Cmax, Cmin) in Subjects During BID Dosing (up to 14 Days Prior to Transitioning to TID Dosing Regimen at PK Visit 1) and up to 35 Days After Transitioning to TID Dosing Regiment (PK Visit 2)
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | PK Visit 1 | PK Visit 2
Number analyzed (Participants) | 13 | 13
ng/mL
  Cmax | 8.60 [1.70 to 18.2] | 8.94 [2.25 to 16.8]
  Cmin | 1.19 [0.290 to 2.50] | 2.14 [0.263 to 6.12]

3. Primary Outcome: To Assess the Pharmacokinetics (AUClast) in Subjects During Twice Daily (BID) Dosing (up to 14 Days Prior to Transitioning to Three Times Daily [TID] Dosing Regimen at PK Visit 1) and up to 35 Days After Transitioning to TID Dosing (at PK Visit 2).
Description: as for outcome 1
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours post-dose at up to 14 days prior to transitioning to TID dosing regimen (PK Visit 1) and at up to 35 days after transitioning to TID dosing regiment (PK Visit 2)
Measure: Mean (Full Range); unit: h*ng/mL
Arm/Group | PK Visit 1 | PK Visit 2
Number analyzed (Participants) | 13 | 13
h*ng/mL | 47.8 [8.92 to 80.6] | 58.0 [10.8 to 109]

4. Secondary Outcome: To Assess 6-minute Walk Distance for Both Groups (BID and TID) 3 to 6 Hours Post-morning Dose.
Description: The 6-minute walk test (6MWT) was conducted at PK Visits 1 and 2, and was performed between hours 3 to 6 post-morning dose to correlate with the predicted peak plasma concentration of oral treprostinil.
Time Frame: The 6MWT was conducted during BID dosing PK collection (up to 14 days prior to transitioning to TID dosing regimen [PK Visit 1]) and during TID dosing PK collection (up to 35 days after transitioning to TID dosing regimen [PK Visit 2]).
Measure: Mean (Full Range); unit: Meters
Arm/Group | PK Visit 1 | PK Visit 2
Number analyzed (Participants) | 13 | 13
Meters | 332.5 [177 to 525] | 347.9 [223 to 541]

5. Secondary Outcome: To Compare the Adverse Event (AE) Profile of BID Versus TID Dosing.
Description: AE diaries including 8 therapy-specific terms were collected during both BID and TID dosing to allow for comparison of events from both regimens. The therapy-specific events included: diarrhea, extremity pain, flushing, headache, hypotension, jaw pain, nausea, and vomiting.
Time Frame: The AEs were recorded for up to 50 days.
Measure: Number; unit: percentage of subjects
Arm/Group | PK Visit 1 | PK Visit 2
Number analyzed (Participants) | 13 | 13
percentage of subjects
  Diarrhea | 46 | 38
  Extremity pain | 54 | 38
  Flushing | 85 | 54
  Headache | 69 | 85
  Hypotension | 23 | 23
  Jaw Pain | 38 | 46
  Nausea | 38 | 77
  Vomiting | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 50 days.
Description: The AEs were recorded by subjects in an AE diary during BID dosing (within 14 days prior to transitioning to TID dosing regimen) and during TID dosing (within 35 days from transition).
Groups:
- PK Visit 1; PK Visit 2: UT-15C SR (treprostinil diethanolamine): open-label study drug
Arm/Group | PK Visit 1 | PK Visit 2
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 13/13 | 13/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PK Visit 1 (N=13) | PK Visit 2 (N=13)
Diarrhea (Gastrointestinal disorders) | 6 (22) | 5 (20)
Extremity pain (Musculoskeletal and connective tissue disorders) | 7 (41) | 5 (47)
Flushing (Vascular disorders) | 11 (57) | 7 (58)
Headache (Nervous system disorders) | 9 (57) | 11 (70)
Hypotension (Vascular disorders) | 3 (8) | 3 (9)
Jaw pain (Musculoskeletal and connective tissue disorders) | 5 (18) | 6 (28)
Nausea (Gastrointestinal disorders) | 5 (31) | 10 (80)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator agree not to publish or publicly present any interim results of the Study without the prior written consent of Sponsor, not to be unreasonably withheld or delayed, except as provided below. Institution and/or Principal Investigator further agree to provide Sponsor with drafts of any such publication or presentation for review and approval no less than 30 days prior to submission for publication or the date of public presentation.